CLINICAL TRIAL: NCT05664126
Title: Haplo-identical Viral-Specific T-cells for Treatment of Cytomegalovirus and Adenovirus Infections After Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VSTHCT; NCI-2023-03240 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cytomegalovirus; Adenovirus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cohort A will include haploidentical donor who is identical to the stem cell donor.
  The first 5 patients will be enrolled in Cohort A. If safety criteria are met, cohort B will be open for enrollment.
  Interventions: Drug: VST infusion; Device: CliniMACS
- Cohort B (Experimental): Cohort B will include haploidentical donor who is different from the stem cell donor
  Interventions: Drug: VST infusion; Device: CliniMACS

INTERVENTIONS:
Drug: VST infusion — single intravenous (IV) infusion.
  Other Names: The product is a suspension of allogenic peripheral blood VSTs enriched based on their secretion of IFN-γ after stimulation with the appropriate antigen
Device: CliniMACS — Cells infusions are prepared using the ClinMACS
  Other Names: ClinMACS Prodigy

SUMMARY:
The investigators want to learn if CMV- and ADV-specific T-cells (cells that fight infections) isolated (selected) from a donor using an automated medical device can be a safe treatment for treating patients with CMV, and ADV after transplant.This study will test the effects and safety of giving VSTs produced here at St. Jude in treating the participant's infection.

Primary objective

To determine the efficacy of VSTs to achieve a ≥1 log10 reduction in CMV and/or ADV viral load in the peripheral blood 4 weeks after VST infusion.

When the initial viral load is <1 log10 above the threshold of detection, the objective is to achieve a reduction to below the threshold of detection.

Secondary objectives

* Determine the safety of VSTs when used to treat CMV and/or ADV viremia post-HCT.
* Determine the proportion of patients who achieve a negative viral load at 3 months post-infusion.
* Assess the persistence of response for 6 months post-infusion.

DETAILED DESCRIPTION:
The study will have 2 cohorts. Cohort A will include haploidentical donor who is identical to the stem cell donor. Cohort B will include haploidentical donor who is different from the stem cell donor. Seropositive donors will be screened for the presence of CMV- and ADV-specific T-cells using a functional flow cytometry assay. The donor will be considered suitable if the percentage of CD3+/IFN-γ+ cells is greater than 0.01% of CD3+ T-cells. Donor leukocytes will be collected using the Spectra Optia system. CMV- and ADV-specific T-cells will be isolated from donor leukocytes by 'IFN-γ-capture' technology using the Prodigy device over a 24-36 hour period and infused.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Patients who have undergone haploidentical HCT or a matched-sibling/matched-unrelated donor HCT, and have CMV and/or ADV detected by PCR in the peripheral blood refractory to antiviral therapy per institutional BMTCT SOP 20.05.
* Definition of "refractory" viremia is persistent positive CMV or ADV viremia after 14 days of treatment per institutional SOP, or an increasing copy number (≥1 log) after 7 days of treatment.
* Patients have no suspected or confirmed GVHD.
* Availability of haploidentical donor for isolation of virus-specific T-cells.
* Have not received a Donor Lymphocyte Infusion in the past 4 weeks.
* Female patients of childbearing age must have a negative pregnancy test.
* Subject, parent, or guardian are capable of giving signed informed consent.
* Patients must have a shortening fraction >26% or left ventricular ejection fraction >40%.
* Patients must have a bilirubin less than or equal to 2.5mg/dL and alanine aminotransferase (ALT) less than or equal to 5 times the upper limit of normal.
* Patients must have an estimated glomerular filtration rate (GFR) greater than 60mL/min/1.73m2 (may use estimated GFR that is auto calculated in the EHR).
* Patients must be free of severe infection which upon determination of the principal investigator precludes therapy with VST.
* Patients must have FVC >50% predicted or able to maintain pulse oximetry saturation > 92% on room air.
* Gut diarrhea <1 liter/day (adults) or <20mL/kg/day (children) or if unable to quantify, then occurrence of 4 stools per day above baseline.
* Patients must have engrafted with an ANC >500 cells/mm3 for 3 consecutive days.

Inclusion criteria for donors

* Age ≥18 years.
* At least single haplotype matched (≥3/6) family member.
* Donor will be identical to the stem cell donor (Cohort A) or different from the stem cell donor (Cohort B).
* HIV negative.
* For females of childbearing age: Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment AND not lactating with intent to breastfeed.
* Regarding donation eligibility, is identified as either having completed the process of donor eligibility determination as outlined in 21CFR 1271 and agency guidance or does not meet 21CFR 1271 eligibility requirements but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21CFR.
* Identified recipient with CMV and/or ADV reactivation post-HCT.

Exclusion Criteria for Patients:

* Active GVHD.
* Pregnancy.
* Inability to provide consent.
* Need for vasopressor or ventilatory support Patients receiving steroids >0.5 mg/kg prednisone equivalent at the time of VST infusion
* Donor Lymphocyte Infusion within 4 weeks prior to VST infusion.
* Receipt of Thymoglobulin or Alemtuzumab within 30 days of VST infusion.
* Other severe uncontrolled concurrent infections (i.e. bacterial or fungal) that are not yet controlled on antimicrobial therapies.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of reduction of CMV and/or ADV viral load | 4 weeks after VST infusion
  The primary objective of this clinical study is to evaluate the efficacy of adoptively transferred CMV- and ADV-specific haploidentical T-cells in patients who have undergone allogeneic HCT. This primary endpoint is defined as ≥1 log10 reduction in CMV and/or ADV viral load 4 weeks after VST infusion. When the initial viral load is <1 log10 above the threshold of detection the endpoint will be a reduction to below the threshold of detection. The success rate will be evaluated using descriptive statistics (sample proportion and standard error). Patients with both CMV and ADC detected will count as success if reduction occurs in one or both of CMV and ADV.

SECONDARY OUTCOMES:
Incidence of infusion-related grade 3-5 adverse events 24 hours after infusion | 24 hours after infusion
  The incidence of infusion-related grade 3-5 adverse events will be estimated using descriptive statistics (sample proportions and cumulative incidence curves with standard errors)
Incidence of AEs related to grade 3-4 cytokine release syndrome (CRS), or grade 1-2 CRS persist beyond 72 hours despite therapy | 4 weeks after VST infusion
  The incidence of AEs related to grade 3-4 cytokine release syndrome (CRS), or grade 1-2 CRS persist beyond 72 hours despite therapy will be estimated using descriptive statistics (sample proportions and cumulative incidence curves with standard errors)
Incidence of Grade 3-4 Neurotoxicity of any duration | 4 weeks after VST infusion
  The incidence of Grade 3-4 Neurotoxicity of any duration will be estimated using descriptive statistics (sample proportions and cumulative incidence curves with standard errors)
Incidence of Grade 3-4 GVHD | 4 weeks after VST infusion
  The incidence of Grade 3-4 GVHD will be estimated using descriptive statistics (sample proportions and cumulative incidence curves with standard errors)
Incidence of grade 3-5 non hematologic toxicities attributable to VST | 4 weeks after VST infusion
  The incidence of grade 3-5 non hematologic toxicities attributable to VST will be estimated using descriptive statistics (sample proportions and cumulative incidence curves with standard errors)
Incidence of secondary graft failure attributable to VST | 4 weeks after VST infusion
  The incidence of secondary graft failure attributable to VST will be estimated using descriptive statistics (sample proportions and cumulative incidence curves with standard errors)
Proportion of patients who achieve a negative viral load result at 3 months | 3 months after VST infusion
  The proportion of patients who achieve a negative viral load result at 3 months will be assessed using descriptive statistics (sample proportions with standard errors)
Persistence of response at 6 months post-infusion | 6 months after VST infusion
  The persistence of response at 6 months post-infusion will be assessed using descriptive statistics (sample proportions with standard errors)

CONTACTS AND LOCATIONS:
Overall Officials: Naik Swati, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St.Jude — http://www.stjude.org/protocols